CLINICAL TRIAL: NCT03126578
Title: Open-label, Single Center, Non-randomized, Fixed Sequence Phase 1 Drug-drug Interaction Study With LEO 32731 and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0058-1324; 2016-003882-24 (EudraCT Number)
Record Dates: First submitted 2017-04-12; First posted 2017-04-24 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-06

CONDITIONS: Drug Interaction Potentiation
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All subjects (Experimental): Part I - Maximum Tolerated Dose: All subjects will receive oral doses of LEO 32731 up-titrated from 10 mg bid on Days 1-3, 20 mg bid on Days 4-6 and 40 mg bid on Days 7-12.
  Part II - Drug-Drug Interaction: All subjects will receive oral doses of LEO 32731 in dose schedule decided upon data from Part I. Subjects will receive a single oral dose of 2.5 mg midazolam on Day -1 prior to the first dose of LEO 32731 and on Days 4, 7 and 17 of multiple dosing with LEO 32731.
  Interventions: Drug: LEO 32731; Drug: Midazolam

INTERVENTIONS:
Drug: LEO 32731 — LEO 32731 is being developed by LEO Pharma.
Drug: Midazolam — Benzodiazepine

SUMMARY:
This is a single center, non-randomized, open-label, fixed sequence study to investigate the effect of multiple oral dosing of LEO 32731 (up-titrated), on CYP3A activity in healthy male subjects using midazolam as a probe CYP3A substrate.

The study will be conducted in two seamless parts:

Part I - Maximal Tolerated Dose (MTD) Part II - Drug-Drug Interaction with midazolam

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will, prior to any study related activities, have given their written informed consent to participate in the study and to abide by the study restrictions.
2. Subjects will be males between 18 and 55 years of age, inclusive.
3. Subjects will have a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive.
4. Subjects must be in good health, as determined by medical history, physical examination, vital signs assessment, 12-lead ECG, and clinical laboratory evaluations.
5. Subjects (including those who have had a vasectomy) must agree to use condoms with spermicide during each sexual intercourse or must agree to be abstinent starting at first drug administration until 3 month after the final dosing.

   Also subjects must agree not to donate sperm in the same time period.
6. Subjects' female partner of childbearing potential must use an additional acceptable method of contraception. Eligible methods are: hormonal contraceptives (oral, injected, implanted, transdermal), intrauterine devices or systems (e.g. hormonal and non-hormonal IUD), barrier methods (condom and diaphragm, condom and cervical cap, etc.) in combination with a spermicide.

Exclusion Criteria:

1. Subjects who have received any prescribed systemic or topical medication within 14 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
2. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration (excluding occasional use of paracetamol or ibuprofen, e.g. in case of pain).
3. Subjects who have received any medications, including St John's Wort known to alter drug absorption or elimination processes (change the enzyme levels) within 30 days of the first dose administration of study drug.
4. Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug with new chemical entity within the past 60 days, or a marketed drug compound within the past 30 days prior to the first dosing.
5. Subjects who have donated any blood, plasma or platelets in 3 months prior to first dosing or who have made donations on more than 3 occasions within the 12 months preceding the first dose administration.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters of midazolam AUC0-t | Day -1 and Day 17
  PK parameters AUC0-t will be analyzed on Day -1 and Day 17.
Pharmacokinetic (PK) parameters of midazolam Cmax | Day -1 and Day 17
  PK parameter Cmax will be analyzed on Day -1 and Day 17.

SECONDARY OUTCOMES:
AUC0-t midazolam | Day 4 and Day 7
  PK parameters of midazolam on Day 4 and Day 7 will only be calculated if relevant differences are seen in midazolam PK parameters between Day -1 and Day 17.
AUC0-inf of midazolam | Day 4 and Day 7
  PK parameters of midazolam on Day 4 and Day 7 will only be calculated if relevant differences are seen in midazolam PK parameters between Day -1 and Day 17.
Cmax of midazolam | Day 4 and Day 7
  PK parameters of midazolam on Day 4 and Day 7 will only be calculated if relevant differences are seen in midazolam PK parameters between Day -1 and Day 17.
AUC0-inf of midazolam | Day -1 and Day 17
  Further PK parameters (AUC0-inf, tmax, t1/2, CL/F and Vz/F) of midazolam on Days -1 and 17 (if applicable these parameters will be calculated on Day 4 and Day 7, too).
Tmax of midazolam | Day -1 and Day 17
  Further PK parameters (AUC0-inf, tmax, t1/2, CL/F and Vz/F) of midazolam on Days -1 and 17 (if applicable these parameters will be calculated on Day 4 and Day 7, too).
t1/2 of midazolam | Day -1 and Day 17
  Further PK parameters (AUC0-inf, tmax, t1/2, CL/F and Vz/F) of midazolam on Days -1 and 17 (if applicable these parameters will be calculated on Day 4 and Day 7, too).
CL/F of midazolam | Day -1 and Day 17
  Further PK parameters (AUC0-inf, tmax, t1/2, CL/F and Vz/F) of midazolam on Days -1 and 17 (if applicable these parameters will be calculated on Day 4 and Day 7, too).
Vz/F of midazolam | Day -1 and Day 17
  Further PK parameters (AUC0-inf, tmax, t1/2, CL/F and Vz/F) of midazolam on Days -1 and 17 (if applicable these parameters will be calculated on Day 4 and Day 7, too).

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Koch, MD, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany